CLINICAL TRIAL: NCT05465330
Title: Effects of Desflurane-propofol Balanced Anesthesia on Visual Evoked Potentials Monitoring: a Randomized Controlled Study
Brief Title: Effects of Desflurane-propofol Balanced Anesthesia on Visual Evoked Potentials Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: wj20220715
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Visual Evoked Potentials
MeSH Terms: interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desflurane Inhalational group (DR group) (Experimental)
  Interventions: Drug: Desflurane
- Desflurane propofol balanced anesthesia group (DPR group) (Active Comparator)
  Interventions: Drug: Desflurane, Propofol

INTERVENTIONS:
Drug: Desflurane — After induction, anesthesia will be maintained with 0.7-1.0 MAC desflurane and remifentanil 0.05-0.2 μg/kg/min
  Arms: Desflurane Inhalational group (DR group)
Drug: Desflurane, Propofol — After induction, anesthesia will be maintained with 0.5 MAC desflurane, propofol 1.5-2.5 μg/ml and remifentanil 0.05-0.2 μg/kg/min
  Arms: Desflurane propofol balanced anesthesia group (DPR group)

SUMMARY:
Intraoperative flash visual evoked potentials (FVEPs) can be used to monitor the integrity of the visual pathway in real-time during surgeries, and is to prevent the damage and deterioration of visual function caused by visual pathway damage, which is the key method of intraoperative monitoring of visual function.

Spinal surgery in the prone position may compress the eyeball and reduce the blood supply of the ophthalmic artery, which is still one of the main causes of postoperative visual impairment. Intraoperative FVEPs monitoring is easily affected by inhale anesthetics, and there is little studies on the effect of intravenous-inhalation balanced anesthesia on FVEPs monitoring. Desflurane wakes up quickly, which is conducive to the recovery of early respiratory function and orientation, and early neurological evaluation. This study aims to compare the effects of desflurane-propofol balanced anesthesia and desflurane pure inhalation anesthesia on the amplitude and latency of FVEPs during spinal surgery under the same sedation depth monitored by bispectral index (BIS) monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing spinal cord surgery under elective general anesthesia;
2. At the same time, other electrophysiological monitoring is required;
3. 18-65 years old;
4. ASA I-III;
5. Sign the informed consent form.

Exclusion Criteria:

1. Patients with visual impairment;
2. Patients with severe liver and kidney function diseases;
3. History of asthma; Uncontrolled hypertension, diabetes, severe arrhythmia or unstable angina pectoris;
4. Have mental illness or unable to communicate;
5. BMI≥30kg/m2；
6. Abuse of analgesics and drug abuse history;
7. Silicone allergy;
8. Visual evoked potential monitoring was rejected.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
N75-p100 amplitude value | 60 minutes after anesthesia induction
  Wave amplitude difference between N75-P100 peak and trough

SECONDARY OUTCOMES:
N75-P100 amplitude decline rates | 30minutes and 60 minutes after anesthesia induction
  The decrease rate of wave amplitude of P100-N145 under corresponding anesthesia maintenance methods compared to the baseline measurements under total intravenous anesthesia
P100-N145 amplitude decline rates | 30minutes and 60 minutes after anesthesia induction
  The decrease rate of wave amplitude of P100-N145 under corresponding anesthesia maintenance methods compared to the baseline measurements under total intravenous anesthesia
P100 latency prolongation rate | 30minutes and 60 minutes after anesthesia induction
  The rate of prolongation of P100 latency compared to the baseline measurements under total intravenous anesthesia
Success rate of FVEP monitoring | 30minutes and 60 minutes after anesthesia induction
  The number of individuals obtaining satisfactory FVEP monitoring waveforms as a ratio to the total number of individuals monitored in each group
FVEPs stacking satisfaction | Intraoperative
  Assessed by the electrophysiological monitoring physician, if good waveforms can be obtained with no more than three superimpositions, it is considered satisfactory
Respiratory recovery time | Within 60 minutes after surgery
  The time from the cessation of anesthesia to the patient's spontaneous breathing recovery
Eye-opening time | Within 60 minutes after surgery
  The time from anesthesia cessation to when the patient can be called to open their eyes
Extubation time | Within 60 minutes after surgery
  The time from the cessation of anesthesia to the removal of the patient's tracheal catheter
Postextubation agitation score | Immediately after extubation, 15 minutes after extubation, 30 minutes after extubation, 1 hour after extubation.
  1 point, calm sleep; 2 points, awake and calm; 3 points, irritable, easily agitated, crying; 4 points, difficult to console, uncontrollable crying; 5 points, unable to settle, confused, delirious.
Ramsay Sedation Score | Immediately after extubation, 15 minutes after extubation, 30 minutes after extubation, 1 hour after extubation.
  1 point - awake, anxious, and restless; 2 points - cooperative, oriented, and calm; 3 points - drowsy, responds to commands; 4 points - drowsy, responds promptly to light tapping on the forehead or loud auditory stimulation; 5 points - drowsy, responds sluggishly to light tapping on the forehead or loud auditory stimulation; 6 points - drowsy, unresponsive. Sedation is considered satisfactory with a score of 2-4, and excessive sedation with a score of 5-6.
Intraoperative anesthetic drugs dosage | The time period between the patient entering the operating room and leaving the operating room
  Including the total amount of intraoperative application of sufentanil, remifentanil, propofol, and rocuronium
Intraoperative vasoactive drugs dosage | The time period between the patient entering the operating room and leaving the operating room
  The total amount of norepinephrine, ephedrine, perdipine, and atropine used during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma J, Wang J, Li Y, Fu Y, Li Y, Qiao H, Han R. Effect of desflurane anesthesia on flash visual evoked potential monitoring in patients undergoing spine surgery: study protocol for a randomized controlled trial. Trials. 2024 Jun 6;25(1):362. doi: 10.1186/s13063-024-08211-9. PMID 38840210